CLINICAL TRIAL: NCT04112121
Title: Hospital-based Ecumenical And Linguistical, Immuno- Neuro-Genetic (HEALING) Study - Randomized Clinical Trial - A Study on the Epigenetic Background of Neuro-immune-modulation in Clinical Environment
Brief Title: Psychological, Neurological and Immunological Changes Following a Meeting With a Chaplain Coupled With Biblical Readings
Acronym: HEALING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr. András Béres, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HEALING STUDY IG/3355/2013
Record Dates: First submitted 2019-09-29; First posted 2019-10-02 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Hospitalism
Keywords: faith; religion; hospitalization; immunology; psychoneuroimmunology; theology; fMRI

STUDY DESIGN:
Intervention Model Description: parallel, randomized, open-labeled, controlled clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients Meeting the Chaplain at the Bedside (Experimental): First meeting with the chaplain, coupled with biblical readings at the bedside.
  Interventions: Behavioral: Meeting with a Chaplain coupled with Biblical Readings
- Patients Meeting the Chaplain at the Chapel (Experimental): First meeting with the chaplain, coupled with biblical readings at the hospital's chapel
  Interventions: Behavioral: Meeting with a Chaplain coupled with Biblical Readings
- Patients Not Meeting the Chaplain (No Intervention): In the control group we enrolled patients whose diagnoses and number of days in the hospital was similar to the intervention groups (covariate-adaptive, blocked, stratified randomization method).

INTERVENTIONS:
Behavioral: Meeting with a Chaplain coupled with Biblical Readings
  Arms: Patients Meeting the Chaplain at the Bedside; Patients Meeting the Chaplain at the Chapel

SUMMARY:
The aim of the "HEALING" " (Hospital-based Ecumenical And Linguistic Immuno-NeuroloGic) Study was to examine immunological and neurological changes in hospitalized participants after meeting a chaplain and Biblical listenings, in order to evaluate whether these meetings affect the course of the disease.

DETAILED DESCRIPTION:
The authors pre-screened hospitalized participants to find those who were the most in need of an intervention by a chaplain. A passage from the Bible was read to the participants during a meeting with the chaplain at the bedside, or in the chapel of the hospital. No meeting occurred in the randomized control group, which was compiled in a way to get a group of participants with an approximatively similar pattern of diagnoses and treatment days than the intervention groups. The pace of enrollment was deliberately slow in order to assure the authenticity of the visits ("slow science"). Blood samples were taken 30 minutes prior, and 60 minutes after the meeting to measure White Blood Cell (WBC)-, lymphocyte counts, interferon gamma (IFN-γ)-, immunoglobulin M (IgM)-, immunoglobulin A (IgA)-, immunoglobulin G (IgG)-, and complement C3 levels. A subgroup of the visited participants was subjected to functional Magnetic Resonance Imaging (fMRI), where they were played an audiotape of readings of the same passage from the Bible. Associative tests, paired-samples t-test, network analysis was performed to search for any correlation between psychological and immunological parameters, completed with Statistical Parametric Mapping to search for correlations of the above with neurological parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult age (>18 years)
* the condition of being hospitalized
* the ability for verbal communication
* alertness, orientation
* no sign of psychosis in their medical history
* willingness to participate in the study after written, informed consent

Exclusion Criteria:

* the inability to communicate verbally
* psychotic state, altered mental state
* unwillingness to participate
* active and treated malignant disease
* steroid, NSAID or metamizole- sodium use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Change in lymphocyte count | Change from baseline at 120 minutes
  lymphocyte count measured with automatised laboratory measurement and microscopic blood smear examination
Change in total white blood cell (WBC) count | Change from baseline at 120 minutes
  WBC count measured with automatised laboratory measurement and microscopic blood smear examination
Change in interferon-gamma level | Change from baseline at 120 minutes
  enzyme-linked immunosorbent assay
Change in immunoglobulin M level | Change from baseline at 120 minutes
  enzyme-linked immunosorbent assay
Change in immunoglobulin A level | Change from baseline at 120 minutes
  enzyme-linked immunosorbent assay
Change in immunoglobulin G level | Change from baseline at 120 minutes
  enzyme-linked immunosorbent assay
Change in complement C3 level | Change from baseline at 120 minutes
  enzyme-linked immunosorbent assay
Change in functional Magnetic Resonance Imaging activity | Change from baseline during the 60 second long activation block
  Statistical Parametric Mapping analysis of Blood Oxygenation Level Dependent (BOLD) answers
Participants' satisfaction with the visit as assessed by Scores given on the "Healing - after" Questionnaire | within 1 hour after intervention
  Participants' assessement of their satisfaction on single-item rating scales in a Questionnaire designed for the Study. Answers range from 1 to 5, with higher values representing better outcomes.
Chaplain's satisfaction with the visit as assessed by Scores given on the "Healing - after" Questionnaire | within 1 hour after intervention
  Chaplain's assessement of her satisfaction on single-item rating scales in a Questionnaire designed for the Study. Answers range from 1 to 5, with higher values representing better outcomes.
Participants' level of distress in the month preceding the measurement as assessed with the total Score of the Perceived Stress Scale 14 (PSS-14) | within 30 minutes before intervention
  PSS-14 Scale uses 14 questions with answers ranging from 0 to 4, with higher values indicating higher levels of distress on the seven negative-, and lower levels of distress on the seven positive items. Scores are obtained by reversing the scores on the seven positive items, then summing across all to give the total PSS-14 Score.
Participants' spiritual and psychological needs, religious practice, thoughts about how they became sick, and how they could heal, as assessed by Scores given on the "Healing - before" Questionnaire | within 30 minutes before intervention
  Participants' assessement on single-item rating scales in a Questionnaire designed for the Study ("Healing - before" Questionnaire). Answers range from 1 to 5, with higher values representing better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: András Béres, M.D., Principal Investigator — Physician
Locations (1):
- Somogy Megyei Kaposi Mór Teaching Hospital, Kaposvár, Hungary

REFERENCES:
- [Derived] Beres A, Emri M, Aranyi C, Fajtai D, Nagy F, Szabo P, Bodecs P, Horcsik E, Perpekne Papp E, Tomanek F, Kuti M, Petofalvine A, Kisdeakne H, Biro G, Kovacs D, Bakos B, Vinczen E, Gal E, Sillinger R, Szalai Z, Szilagyi A, Kiss-Merki M, Nagyeri G, Fodor J, Nemeth T, Papp E, Repa I. Healing through faith: Meeting a chaplain coupled with biblical readings could produce lymphocyte changes that correlate with brain activity (HEALING study). F1000Res. 2024 Oct 30;10:1295. doi: 10.12688/f1000research.74504.5. eCollection 2021. PMID 40496603